CLINICAL TRIAL: NCT00588952
Title: NMDA Dysregulation in Individuals With a Family Vulnerability to Alcoholism
Brief Title: Ketamine/Placebo Family History Positive Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0103012310; VA Alcohol Research Center (Other Grant/Funding Number: VA Alcohol Research Center Grant); P50AA012870 (NIH)
Record Dates: First submitted 2007-12-27; First posted 2008-01-09 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family History Positive (Experimental): Subjects with a positive family history of alcoholism
  Interventions: Drug: Ketamine and Placebo
- Family History Negative (Experimental): Subjects with a negative family history of alcoholism
  Interventions: Drug: Ketamine and Placebo

INTERVENTIONS:
Drug: Ketamine and Placebo — Two test days will involve administration of placebo and Ketamine (0.23 mg/kg, loading dose and infusion rate 0.58 mg/kg/minute) intravenously for 60 minutes
  Other Names: intravenous

SUMMARY:
The proposed study is the first to explore the contribution of brain glutamate systems, a major target of ethanol in the brain, to the vulnerability to develop alcoholism. This study may lead to an enhanced understanding of the underlying neurobiological mechanism in high-risk individuals that may lead to the transition from moderate to excessive use of alcohol.

DETAILED DESCRIPTION:
Males and females with a paternal family history of alcoholism have a high risk for developing alcoholism. These individuals have been shown to decrease dysphoric responses to alcohol self-administration that may promote the excessive use of alcohol. Ethanol has been shown to be an antagonist at the N-methyl-D-aspartate (NMDA) glutamate receptor. We have recently shown that sober alcoholics have decreased dysphoric response to the NMDA antagonist, ketamine. We propose to test the hypothesis that this characteristic exists as a vulnerability factor in those individuals susceptible to develop alcoholism. Specifically, the objective is to determine whether individuals with a family history positive (FHP) for alcoholism will experience less dysphoric, anxiogenic, and psychotogenic effects to ketamine infusion when compared to family history negative (FHN) control subjects.

Male and female subjects, FHP (biological father and one other first degree relative) between the ages of 21-30, and matched controls (FHN) will complete 2 test days in a randomized balanced order under double-blind conditions. Test days will involve the 60-minute intravenous infusion of placebo and ketamine. Outcome measures include the Biphasic Alcohol Scale and visual analog scales for mood states. Secondary measures include visual analog scales for high, similarity to ethanol, the Sensation Scale (a validated measure of ethanol-like sensations) and aspects of craving for alcohol.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female between the ages of 21 and 30 years
2. Medically and neurologically healthy on the basis of history, physical examination, EKG, screening laboratories, absence of current and/or past substance abuse

For Family History Positive (FHP) Subjects: Biological father and another first or second-degree biological relative with history of alcoholism

Exclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) psychiatric and substance abuse diagnosis by history on psychiatric evaluation that includes a structured diagnostic interview (The Semi-Structured Assessment for the Genetics of alcoholism: SSAGA) and the Wisconsin Scales of Psychosis Proneness
2. History of counseling or psychotherapy; except family therapy centered around another family member
3. Extended unwillingness to remain alcohol-free for three days prior to testing and for the duration of the testing period
4. For women: positive pregnancy test at screening or intention to engage in unprotected sex during the study
5. Alcohol naïve
6. Previous bad experience with ketamine
7. Adoptee and no contact with family members

For Family History Negative (FHN) Subjects: NO family history of alcoholism in any first or second-degree relatives (subjects must reliably report on three first-degree relatives)

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2001-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L. Petrakis, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Background] Yoon G, Pittman B, Limoncelli D, Krystal JH, Petrakis IL. Familial Alcoholism Risk and the Ratio of Stimulant to Sedative Effects of Ketamine. Biol Psychiatry. 2016 May 1;79(9):e69-e70. doi: 10.1016/j.biopsych.2015.09.006. Epub 2015 Sep 25. No abstract available. PMID 26475672

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Family History Positive | Family History Negative
Started | 29 | 70
Completed | 26 | 63
Not Completed | 3 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Population: All available data was utilized in the analysis using mixed models
Groups:
- Total: Total of all reporting groups
Arm/Group | Family History Positive | Family History Negative | Total
Number analyzed (Participants) | 29 | 70 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 70 | 99
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.97 (3.02) | 24.13 (2.34) | 24.37 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 36 | 49
  Male | 16 | 34 | 50
Region of Enrollment [Number; unit: participants]
  United States | 29 | 70 | 99

OUTCOME MEASURES:

1. Primary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedation
Description: Self-reporting rating scale to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol effects. We used the BAES to measure alcohol-like effects in subjects that received ketamine infusions.
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family History Positive: Subjects with a positive family history of alcoholism
  Ketamine: Ketamine: 0.23 mg/kg, loading dose and infusion rate 0.58 mg/kg/minute for 60 minutes, IV
  Placebo: Placebo: loading dose and an infusion for 60 minutes saline solution
- Family History Negative: Subjects with a negative family history of alcoholism
  Ketamine: Ketamine: 0.23 mg/kg, loading dose and infusion rate 0.58 mg/kg/minute for 60 minutes, IV
  Placebo: Placebo: loading dose and an infusion for 60 minutes saline solution
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 29 | 70
units on a scale
  Ketamine: number analyzed (Participants) | 27 | 68
  Ketamine | 0.63 (1.15) | 0.96 (2.14)
  Placebo: number analyzed (Participants) | 28 | 65
  Placebo | 0.71 (2.18) | 1.25 (2.46)

2. Primary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedation
Description: as for outcome 1
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 29 | 70
units on a scale
  Ketamine: number analyzed (Participants) | 26 | 66
  Ketamine | 18.96 (14.92) | 24.74 (17.34)
  Placebo: number analyzed (Participants) | 28 | 66
  Placebo | 2.46 (7.12) | 1.36 (2.89)

3. Primary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedation
Description: as for outcome 1
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 29 | 70
units on a scale
  Ketamine: number analyzed (Participants) | 25 | 66
  Ketamine | 18.36 (12.49) | 25.06 (18.22)
  Placebo: number analyzed (Participants) | 28 | 66
  Placebo | 1.46 (4.34) | 1.64 (4.03)

4. Primary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedation
Description: as for outcome 1
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 29 | 70
units on a scale
  Ketamine: number analyzed (Participants) | 26 | 65
  Ketamine | 7.46 (12.16) | 9.99 (13.04)
  Placebo: number analyzed (Participants) | 28 | 66
  Placebo | 1.07 (3.16) | 0.92 (2.03)

5. Primary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulation
Description: Self-reporting rating scale to measure the stimulation effects (0 not at all stimulated - 70 extremely stimulated) of alcohol effects. We used the BAES to measure alcohol-like effects in subjects that received ketamine infusions.
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 29 | 70
units on a scale
  Ketamine: number analyzed (Participants) | 27 | 68
  Ketamine | 3.78 (8.66) | 2.43 (7.25)
  Placebo: number analyzed (Participants) | 28 | 66
  Placebo | 2.36 (6.14) | 2.88 (7.57)

6. Primary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulation
Description: as for outcome 5
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 29 | 70
units on a scale
  Ketamine: number analyzed (Participants) | 26 | 66
  Ketamine | 22.39 (22.53) | 14.58 (15.72)
  Placebo: number analyzed (Participants) | 28 | 66
  Placebo | 1.82 (4.10) | 1.82 (5.5)

7. Primary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulation
Description: as for outcome 5
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 29 | 70
units on a scale
  Ketamine: number analyzed (Participants) | 25 | 66
  Ketamine | 15.4 (19.09) | 9.06 (12.69)
  Placebo: number analyzed (Participants) | 28 | 66
  Placebo | 1.54 (3.50) | 1.64 (5.29)

8. Primary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulation
Description: as for outcome 5
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 29 | 70
units on a scale
  Ketamine: number analyzed (Participants) | 26 | 65
  Ketamine | 3.81 (8.45) | 3.02 (8.12)
  Placebo: number analyzed (Participants) | 28 | 66
  Placebo | 1.61 (3.66) | 2.12 (6.42)

ADVERSE EVENTS:
Arm/Group | Family History Positive | Family History Negative
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/70
Other Adverse Events (participants affected / at risk) | 0/29 | 2/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family History Positive (N=29) | Family History Negative (N=70)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — Subjects stopped infusion felt very anxious
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject vomited during infusion so infusion was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes